CLINICAL TRIAL: NCT05560568
Title: Effects of Optimizing Nocturnal Glycemic Control on Sleep Parameters in Type 1 Diabetes
Acronym: DIABNIGHT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0533
Record Dates: First submitted 2022-09-22; First posted 2022-09-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes, Sleep, nocturnal glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with type 1 diabetes: Adult patients with type 1 diabetes treated with insulin pumps according to current recommendations with an indication to switch to a hybrid closed-loop pump
  Interventions: Other: Sleep parameters data collection

INTERVENTIONS:
Other: Sleep parameters data collection — Sleep parameters collected before and after hybrid close-loop pump activation. Data collected with adequate devices (i.e. actigraph and Dreem Band).

SUMMARY:
Sleep is crucial for physical and mental health. Environmental, social, or professional pressures can cause sleep duration to fall below the recommended 7-9 hours of sleep per night. Young adults with type 1 diabetes, have additional interference with fear, control and management of hypo/hyperglycemia management, alarms from their devices, which delay bedtime, disrupt sleep and generate multiple awakenings and difficulty returning to sleep. Sleep disturbance is correlated with blood glucose variability as recently demonstrated by a coupled analysis of sleep and glucose level collected by Continuous Glucose Monitoring (CGM). In this study, higher glucose variability predicted impaired sleep at the individual level.

Automated insulin infusion has shown impressive results in clinical and real-life studies, with more than 90% of patients achieving good glycemic control. Il seems to improve sleep quality in subjects after 4 weeks in hybrid closed-loop, self-administered studies compared to a control group.

The main objective of our study is to measure the positive influence of a better glycemic control on the different sleep parameters in subjects with type 1 diabetes at the time of the passage in hybrid closed-loop and in comparison to an identical period in open-loop.

ELIGIBILITY:
Inclusion Criteria:

* Patients usually followed by the Diab-eCare service (HCL), male or female, between 18 and 50 years old,
* Confirmed diagnosis of type 1 diabetes for more than 1 year regardless of age of diagnosis,
* Eligible according to current recommendations and the center's practices for a hybrid closed-loop solution including all Dexcom G6,
* On pump, whatever the device used, for at least 6 months and with a Dexcom G6 CGM sensor for at least one month with more than 95% of data obtained,
* BMI<30 kg/m2,
* HbA1C <10%,
* Do not oppose to the said research.

Exclusion Criteria:

* Patients with type 2 diabetes,
* Patients with a cause other than diabetes that could disrupt sleep:

  * Known or suspected sleep apnea syndrome with high risk according to the Berlin questionnaire, And/or
  * Presence of risk factors such as severe retinopathy, nephropathy, hypertension, autonomic neuropathy, chronic psychiatric disorders, endocrine or metabolic pathologies that have not been stabilized, therapeutics that may alter sleep (i.e. sleeping pills, corticosteroids, antidepressants, anxiolytics, antihistamines), regular use of cannabis, abusive use of alcohol (regularly > 3 drinks per day for a man and > 2 drinks for a woman) And/or
  * Night or shift work,
* Inability to collect data and/or understand the objectives of the study according to the investigator,
* Persons under legal protection,
* Persons not affiliated with a social security system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 20 adult patients with type 1 diabetes with an indication to switch to a hybrid closed-loop pump according to current recommendations. They will be informed of the study during a routine consultation at the Diab-eCare unit (Hospices Civils of Lyon, Lyon, France).
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | Change between inclusion and 1 month after the switch to the hybrid closed loop
  To evaluate if the optimization of glycemic control after 1 month of use of a hybrid closed loop improves sleep efficiency, i.e. the change of ratio of measured sleep time to time in bed * 100, evaluated by the actiwatch 2 (AW2) actigraph from inclusion (before the switch to the hybrid closed loop) to 1 month after the switch.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre du diabète Diab-eCare, Lyon, France